CLINICAL TRIAL: NCT03379285
Title: Risk Factors for Further Bleeding in Patients Admitted to Intensive Care for Gastro Intestinal Bleeding
Brief Title: Management of Digestive Haemorrhaging In CHRU of Brest During 2009 and 2014
Acronym: HDréa
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: HDréa
Record Dates: First submitted 2017-11-23; First posted 2017-12-20 (Actual); Last update posted 2017-12-20 (Actual); Status verified 2017-10

CONDITIONS: Gastro Intestinal Bleeding
Keywords: Gastro Intestinal Bleeding;; Transfusion,; Outcomes
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Gastro intestinal (GI) bleeding is relatively frequent and may lead to intensive care unit admission. Although a restrictive strategy for red blood cell transfusion is supported by a large randomized controlled trial literature, less is known about the impact of transfusion strategy of other blood components and administration of anti fibrinolytic on clinical outcomes.

This study aims to identify parameters that may be associated with the risk of further bleeding in patients admitted to ICU for GI bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Gastro Intestinal Bleeding admitted to either medical or surgical intensive care unit

Exclusion Criteria:

* patients retrieved from another hospital
* age < 18 years consent withdrawal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to intensive care unit with the primary admission diagnosis of Gastro Intestinal Bleeding and who were not retrieved from another hospital.
Sampling Method: Non-Probability Sample
Enrollment: 272 (Actual)
Dates: Start 2016-10-03 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Bleeding | within a week
  Bleeding persistance or recidive requiring an intervention or a scope

SECONDARY OUTCOMES:
mortality | during hospitalisation (28 days)
  hospital mortality

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France